CLINICAL TRIAL: NCT02619279
Title: A Livelihood Intervention for Impoverished Women and Children in Rural Uganda: Randomized Controlled Trial
Brief Title: A Livelihood Intervention for Impoverished Women and Children in Rural Uganda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other)
Responsible Party: Principal Investigator, Alexander Tsai, Assistant Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MH096620-S4
Record Dates: First submitted 2015-08-15; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Indigency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate treatment (Experimental): Participants' mothers will receive a livelihood intervention package consisting of a orientation and training and a loan package of chickens and associated implements to create poultry microenterprises
  Interventions: Other: Livelihood intervention
- Delayed treatment (No Intervention): Participants' mothers will receive no intervention but will be placed on a waitlist to receive the intervention after a 12-month delay.

INTERVENTIONS:
Other: Livelihood intervention — Participants' mothers will receive a livelihood intervention package consisting of a orientation and training and a loan package of chickens and associated implements to create poultry microenterprises.
  Arms: Immediate treatment

SUMMARY:
The objective of the study is to determine whether a livelihood intervention can improve health and schooling outcomes of the children of woman participating in a livelihood intervention in rural Uganda.

ELIGIBILITY:
Inclusion Criteria:

* All children under 18 years

Exclusion Criteria:

* Adults older than 18 years

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Stunting based on Anthropometric Measurements | 12 months
  Height-for-age calculated based on child height and child age, measured for children under 5 years of age
Weight-for-Height based on Anthropometric Measurements | 12 months
  Weight-for-height calculated based on child height and child weight, measured for children under 5 years of age
Raven's Colored Progressive Matrices test | 12 months
  Raven's Colored Progressive Matrices test score (range, 0-18), measured for children aged 5-8 years
Mullen Early Learning Scales | 12 months
  Mullen Early Learning Scales: 144 items total, divided across 4 subtests in visual receptive organization, visual expressive organization, language expressive organization, and language receptive organization
Home Observation of the Measurement of Environment Scale | 12 months
  Home Observation of the Measurement of Environment, modified for the Ugandan context (58 items distributed across the following domains: Responsivity, Encouragement of maturity, Emotional climate, Learning materials and opportunities, Enrichment, Family companionship, Family integration and Physical environment)

SECONDARY OUTCOMES:
Child Educational Investment Scale | 12 months
  Average time spent on school and schoolwork in the past 7 days (number of hours)
Child Non-Educational Investment Scale | 12 months
  Average time spent on household chores and playing in the past 7 days (number of hours)
Mother's Educational Investment Scale | 12 months
  Average time spent on reading to children or helping with homework in past 7 days (number of hours)
Mother's Aspirations for Child Education Scale | 12 months
  Mother's aspiration for child's educational attainment, ranging from 1 (finish P7 primary school) to 5 (finish graduate school)
Mother's Aspirations for Child Career Scale | 12 months
  Mother's aspirations for child's adult employment by age 25 (with the option to select one of 33 different blue-collar and white-collar occupational categories)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Tsai, MD, PhD, Principal Investigator — Massachusetts General Hospital; Bernard Kakuhikire, MBA, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda